CLINICAL TRIAL: NCT00616785
Title: Phase II Trial Irinotecan and Cisplatin Induction Chemotherapy Followed by Radiotherapy Concurrently With Etoposide/Cisplatin in Locally Advanced, Unresectable Stage III Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Stage III Non-Small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000584442; YONSEI-4-2007-0120
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2008-09

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Etoposide; Irinotecan; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Drug: irinotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, cisplatin, and etoposide work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving combination chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with radiation therapy works in treating patients with stage III non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of induction chemotherapy comprising irinotecan hydrochloride and cisplatin in patients with locally advanced, unresectable stage III non-small cell lung cancer.
* To evaluate the feasibility of radiotherapy administered concurrently with etoposide and cisplatin chemotherapy after induction chemotherapy in these patients.

Secondary

* To evaluate the toxicity of induction chemotherapy comprising irinotecan hydrochloride and cisplatin in these patients.
* To assess whether this induction chemotherapy regimen will improve patient survival when compared with outcomes from the predecessor study, SWOG-9019.

OUTLINE: Patients receive dose-dense induction chemotherapy comprising irinotecan hydrochloride IV and cisplatin IV on days 1 and 8. Treatment repeats every 21 days for up to 2 courses.

After completion of induction chemotherapy, patients undergo radiotherapy five days a week for approximately 7 weeks. Patients receive concurrent chemotherapy comprising cisplatin IV on days 1, 8, 29, and 36 and etoposide IV on days 1-5 and 29-33.

After completion of study therapy, patients are followed at 6 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIA (N2) or IIIB disease

    * Pathologic documentation of N2-3 mediastinal lymph nodes is encouraged but not required if nodal size is ≥ 1.5 cm in largest diameter
    * No stage IIIB disease with malignant pleural effusion or superior sulcus tumor
* At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors
* Unresectable disease
* No known brain metastasis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* ANC ≥ 1,500/mm³
* Hemoglobin ≥ 9.0 g/dL (can be corrected by transfusion)
* Platelet count ≥ 100,000/mm³
* Creatinine < 1.5 mg/dL
* Total bilirubin < 2 times upper limit of normal (ULN)
* Transaminases < 3 times ULN
* Patient compliance and geographic proximity that allow adequate follow up
* No serious, uncontrolled systemic intercurrent illness (e.g., infections or poorly controlled diabetes)
* No history of significant neurological or mental disorder, including seizures or dementia
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanoma skin cancer
* No active cardiac disease not controlled by therapy
* No myocardial infarction within the past 12 months

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for NSCLC
* No other concurrent systemic chemotherapy, investigational drug, or radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Rate of local/regional control
Rate of systemic disease control
Feasibility of radiotherapy administered concurrently with etoposide and cisplatin chemotherapy

SECONDARY OUTCOMES:
Toxicity of irinotecan hydrochloride and cisplatin induction chemotherapy as assessed by NCI CTCAE v3.0
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hang Kim, MD, Study Chair — Yonsei University
Locations (1):
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea